CLINICAL TRIAL: NCT04460742
Title: CAPABLE Transitions: A Randomized, Unblinded, 60-Subject Clinical Trial of an Occupational Therapy-Led In-Home Intervention to Help Older Adults Transition to Their Homes Following Hospital or Post-Acute Care Facility Discharge
Brief Title: CAPABLE Transitions: A Home Health-Based Intervention for the Hospital or Post-Acute Care Facility-to-Home Transition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Adam Simning, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00004519; 5K23AG058757-02 (NIH); 3 K 23 AG058757-02S1 (Other Grant/Funding Number: National Institute of Aging)
Record Dates: First submitted 2020-06-26; First posted 2020-07-08 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Care Transitions; Dementia
Keywords: Post-acute care; Home health agency
MeSH Terms: conditions — Dementia | interventions — Home Care Agencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAPABLE Transitions (Experimental): Older adults admitted to University of Rochester Medicine Home Care with and without dementia will receive care as usual as well as CAPABLE-trained occupational therapy, registered nurse, and handyman services delivered over 3-4 months.
  Interventions: Behavioral: CAPABLE Transitions; Behavioral: Home Health Agency Care
- Care As Usual (Active Comparator): Older adults admitted to University of Rochester Medicine Home Care (a Medicare-certified home health agency) with and without dementia will receive care as usual.
  Interventions: Behavioral: Home Health Agency Care

INTERVENTIONS:
Behavioral: CAPABLE Transitions — The CAPABLE Transitions intervention group will receive an occupational therapy-led multidisciplinary in-home intervention in which the study occupational therapist (<6 visits), registered nurse (<5 visits), and handyman (<2 visits) work with participants over 3-4 months. This intervention group also will receive home health agency care as usual services. CAPABLE Transitions in embedded within a home health agency and includes a care transitions emphasis.
  Arms: CAPABLE Transitions
Behavioral: Home Health Agency Care — Both the CAPABLE Transitions intervention and care as usual treatment arms will receive home health agency care as usual services, which can include nursing, health aide, medical social work, and occupational, physical, and speech therapy services. Home health agency clinicians will determine the types and duration of CHHA services that the study participants receive; these services will be completely independent from the research study.

SUMMARY:
This clinical study is designed to test the feasibility of a new intervention, CAPABLE Transitions. CAPABLE Transitions is based on the Community Aging in Place, Advancing Better Living for Elders (CAPABLE) intervention designed by Dr. Sarah Szanton at Johns Hopkins University. Similar to CAPABLE, CAPABLE Transitions consists of an occupational therapy (OT)-led intervention in which the study OT, nurse, and handyman deliver an in-home intervention over 3-4 months. This intervention is designed to help with the transition of care from a hospital or post-acute care facility discharge as well as to optimize functioning and home safety. This clinical study plans to recruit a total of 60 older adults with and without dementia admitted to a home health agency following discharge from a hospital or post-acute care facility. Given that this is a feasibility study, it is not designed or powered to test hypotheses.

DETAILED DESCRIPTION:
This pilot study is a randomized, care-as-usual (CAU)-comparator, unblinded clinical trial of an occupational therapy (OT)-led in-home intervention designed to help older adults successfully return to and remain in their homes following discharge from a hospital or post-acute care facility (e.g., skilled nursing or inpatient rehabilitation facilities). This intervention is called CAPABLE Transitions. In total, 60 adults (36 in the intervention arm, 24 in the CAU arm) aged 65 years and older recently discharged from a hospital or post-acute care facility and admitted to a Medicare-certified home health agency (CHHA) with and without dementia will be recruited. This pilot study's main outcomes relate to the feasibility of the study. These outcomes include study recruitment and retention, fidelity to and perceived benefit of the intervention, and data completeness with regard to clinical outcomes (e.g., home time, quality of life, and health care utilization).

This study will recruit English-speaking adults aged 65 years and older who live in the Rochester region and are admitted to a CHHA following a hospital or post-acute care facility stay. There are two treatment groups. The intervention group will receive CAPABLE Transitions as well as CHHA CAU services. The CAU group will receive CHHA CAU services, which can include nursing, health aide, medical social work, and occupational, physical, and speech therapy services. CHHA clinicians will determine the types and duration of CHHA services that the study participants receive; these services will be completely independent from the research study.

Assessment interviews will be conducted at baseline as well as at three and six month follow-up. Interviews will assess sociodemographics, health and functioning, mental health and cognitive functioning, home environment, medical services use, and intervention feedback. Information also will be extracted on medical conditions, medications, communication with providers, and services utilization from participants' medical records.

ELIGIBILITY:
Inclusion Criteria:

* admitted to Medicare-certified home health agency following discharge from a hospital, inpatient rehabilitation facility, or skilled nursing facility
* live in Rochester, NY region
* aged 65 years or older
* English-speaking

Exclusion Criteria:

* plan to move within one year
* has a terminal diagnosis (e.g., < 1-year life expectancy, in hospice)
* receiving active cancer treatment (active treatment includes surgery or a course of radiation or chemotherapy; it does not include long-term maintenance treatment such as daily hormonal treatment of prostate cancer)
* inability or unwillingness of individual or legal guardian/representative to give written informed consent or assent
* has been discharged from a hospital or post-acute care facility for more than 28 days
* are COVID-19 positive, have suspected COVID-19 infection, or resides with a person who is COVID-19 positive or has suspected COVID-19

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Simning, MD, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon request as part of a academic collaboration

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CAPABLE Transitions | Care As Usual
Started | 16 | 15
Completed | 14 | 14
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CAPABLE Transitions | Care As Usual | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 77 (6.66) | 71.8 (6.33) | 74.5 (6.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 15 | 14 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 0 | 2
  White | 12 | 15 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Screened as Eligible
Description: The study will monitor how many older adults are screened and satisfy the eligibility criteria.
Time Frame: For each potential participant, this outcome is determined prior to possible study enrollment.
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study Screening and Recruitment: This section refers to all of the people screened and ultimately recruited into the study, prior to randomization to different treatment arms.
Arm/Group | Overall Study Screening and Recruitment
Number analyzed (Participants) | 311
Participants | 180

2. Primary Outcome: Percentage of Screened Participants That Enroll
Description: The study will monitor how many older adults who satisfy the eligibility criteria are enrolled in the study.
Time Frame: This outcome is determined at the time of study enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Screening and Recruitment
Number analyzed (Participants) | 180
Participants | 31

3. Primary Outcome: Percentage of Enrolled Participants That Are Retained
Description: The study will monitor the percentage of participants that complete the study.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CAPABLE Transitions | Care As Usual
Number analyzed (Participants) | 16 | 15
Participants | 14 | 14

4. Primary Outcome: Percentage of Participants Who Perceive a Benefit From the Intervention
Description: Participants and study partners will be asked Likert-item response survey questions to assess the perceived benefit and burdensomeness of the intervention.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | CAPABLE Transitions
Number analyzed (Participants) | 14
Participants | 13

5. Primary Outcome: Percentage of Participants Who Perceive a Benefit From the Intervention
Description: as for outcome 4
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CAPABLE Transitions
Number analyzed (Participants) | 13
Participants | 12

6. Primary Outcome: Proportion of Critical Tasks Completed
Description: The study will review audio recordings and study interventionists' documentation to examine fidelity to the intervention and score whether the interventionists completed the central tasks of CAPABLE Transitions. The study will score completion of the critical components as "yes" or "no" and this outcome will be reported as the proportion of critical components of the CAPABLE Transitions intervention that were completed by the occupational therapist and registered nurse.
Time Frame: Throughout Study Intervention, an average of 5 months
Measure: Mean (Standard Deviation); unit: Proportion of Critical Tasks Completed
Units Other Than Participants: Critical Tasks
Arm/Group | CAPABLE Transitions
Number analyzed (Participants) | 16
Number analyzed (Critical Tasks) | 40
Proportion of Critical Tasks Completed | 0.89 (0.08)

7. Primary Outcome: Data Completeness on Clinical Outcomes
Description: The study will monitor the percentage of participants who have complete information on home time, quality of life, and health services utilization at 3 months.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | CAPABLE Transitions | Care As Usual
Number analyzed (Participants) | 16 | 15
Participants | 16 | 14

8. Primary Outcome: Data Completeness on Clinical Outcomes
Description: The study will monitor the percentage of participants who have complete information on home time, quality of life, and health services utilization at 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CAPABLE Transitions | Care As Usual
Number analyzed (Participants) | 16 | 15
Participants | 14 | 13

9. Secondary Outcome: Home Time in Days (From the Baseline to 3 Month Period)
Description: Home time is the number of days participants spend alive in non-institutional settings (e.g., nursing homes and hospitals). The study will report the participants' home time from baseline to 3 months of follow-up.
Time Frame: Baseline to Month 3 (3 months)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CAPABLE Transitions | Care As Usual
Number analyzed (Participants) | 16 | 15
days | 87.94 (7.25) | 88.67 (3.99)

10. Secondary Outcome: Home Time in Days (From the 3 to 6 Month Period)
Description: Home time is the number of days participants spend alive in non-institutional settings (e.g., nursing homes and hospitals). The study will report the participants' home time from 3 to 6 months of follow-up.
Time Frame: Month 3 to Month 6 (3 months)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CAPABLE Transitions | Care As Usual
Number analyzed (Participants) | 16 | 14
days | 89.38 (2.00) | 89.86 (0.36)

11. Secondary Outcome: Mean Change in Quality of Life Using EQ-5D-5L (Unabbreviated Title)
Description: The study will examine quality of life (EQ-5D-5L) among study participants at 3 months of follow-up (positive scores indicate improvement from baseline).
  Rating: mobility, self-care, usual activities, pain/discomfort and anxiety/depression, each with 1 as lowest score and 5 as highest score: no problems, slight problems, moderate problems, severe problems and extreme problems, where higher scores indicate worse outcome.
  The EQ VAS question records the patient's self-rated health on a vertical visual analogue scale from 0 to 100, where the endpoints are labelled 'The best health you can imagine' (score=100) and 'The worst health you can imagine' (score=0). Therefore higher scores may indicate better outcomes.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAPABLE Transitions | Care As Usual
Number analyzed (Participants) | 15 | 14
score on a scale
  Mobility Change | 0.73 (1.33) | 1.07 (1.07)
  Self-Care Change | 0.40 (0.74) | 0.50 (0.76)
  Usual Activities Change | 0.73 (1.39) | 0.79 (1.05)
  Pain/Discomfort Change | -0.07 (0.96) | 0.36 (1.50)
  Anxiety/Depression Change | -0.13 (0.64) | 0.14 (0.77)
  Self-Rated Health Change | 6.27 (28.29) | 1.43 (15.80)

12. Secondary Outcome: Mean Change in Quality of Life Using EQ-5D-5L (Unabbreviated Title)
Description: The study will examine quality of life (EQ-5D-5L) among study participants at 6 months of follow-up (positive scores indicate improvement from baseline).
  Rating: mobility, self-care, usual activities, pain/discomfort and anxiety/depression, each with 1 as lowest score and 5 as highest score: no problems, slight problems, moderate problems, severe problems and extreme problems, where higher scores indicate worse outcome.
  The EQ VAS question records the patient's self-rated health on a vertical visual analogue scale from 0 to 100, where the endpoints are labelled 'The best health you can imagine' (score=100) and 'The worst health you can imagine' (score=0). Therefore higher scores may indicate better outcomes.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CAPABLE Transitions | Care As Usual
Number analyzed (Participants) | 14 | 14
score on a scale
  Mobility Change | 0.57 (1.09) | 0.71 (1.07)
  Self-Care Change | 0.50 (0.94) | 0.36 (0.93)
  Usual Activities Change | 1.21 (1.19) | 0.93 (1.07)
  Pain/Discomfort Change | 0.29 (1.07) | 0.50 (1.40)
  Anxiety/Depression Change | -0.36 (1.01) | -0.29 (0.73)
  Self-Rated Health Change | 8.07 (26.83) | 10.5 (12.91)

13. Secondary Outcome: Health Services Use, Percentage
Description: The study will examine the percentage of participants who went to the emergency department, were hospitalized, and were admitted to a skilled nursing facility from baseline to 3 months of follow-up.
Time Frame: Baseline to Month 3 (3 months)
Measure: Count of Participants; unit: Participants
Arm/Group | CAPABLE Transitions | Care As Usual
Number analyzed (Participants) | 16 | 15
Participants
  ED Visit | 1 | 1
  Hospitalization | 2 | 2
  Skilled Nursing Facility Admission | 0 | 0

14. Secondary Outcome: Health Services Use, Percentage
Description: The study will examine the percentage of participants who went to the emergency department, were hospitalized, and were admitted to a skilled nursing facility from 3 to 6 months of follow-up.
Time Frame: Month 3 to Month 6 (3 months)
Measure: Count of Participants; unit: Participants
Arm/Group | CAPABLE Transitions | Care As Usual
Number analyzed (Participants) | 16 | 14
Participants
  ED Visit | 3 | 2
  Hospitalization | 2 | 0
  Skilled Nursing Facility Admission | 0 | 0

15. Secondary Outcome: Health Services Use, Mean
Description: The study will tabulate the mean number of times participants went to the emergency department, were hospitalized, and were admitted to a skilled nursing facility from baseline to 3 months of follow-up.
Time Frame: Baseline to Month 3 (3 months)
Measure: Mean (Standard Deviation); unit: events
Arm/Group | CAPABLE Transitions | Care As Usual
Number analyzed (Participants) | 16 | 15
events
  ED Visit | 0.06 (0.25) | 0.07 (0.26)
  Hospitalization | 0.13 (0.34) | 0.27 (0.70)
  Skilled Nursing Facility Admission | 0 (0) | 0 (0)

16. Secondary Outcome: Health Services Use, Mean
Description: The study will tabulate the mean number of times participants went to the emergency department, were hospitalized, and were admitted to a skilled nursing facility from 3 to 6 months of follow-up.
Time Frame: Month 3 to Month 6 (3 months)
Measure: Mean (Standard Deviation); unit: events
Arm/Group | CAPABLE Transitions | Care As Usual
Number analyzed (Participants) | 16 | 14
events
  ED Visit | 0.19 (0.40) | 0.14 (0.73)
  Hospitalization | 0.13 (0.34) | 0 (0)
  Skilled Nursing Facility Admission | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: From study recruitment to termination of data collection, an average of 6 months.
Description: At every study visit, study interventionists and research coordinators asked about any medical events that occurred since the prior visit. We also reviewed the participants' medical charts at 3 and 6 months, which provided information about medical events. Of note, none of the serious adverse events were believed to be study related.
Arm/Group | CAPABLE Transitions | Care As Usual
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 5/16 | 1/15
Other Adverse Events (participants affected / at risk) | 3/16 | 1/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CAPABLE Transitions (N=16) | Care As Usual (N=15)
Muscle cramping or swelling (Musculoskeletal and connective tissue disorders) | 1 | 1
Abdominal pain and discomfort (Gastrointestinal disorders) | 2 | 1
Fall with injury (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint infection (Infections and infestations) | 1 | 0
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Substance intoxication (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CAPABLE Transitions (N=16) | Care As Usual (N=15)
Fall (Metabolism and nutrition disorders) | 0 | 1
Minor back fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
COVID-19 Exposure (Infections and infestations) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/42/NCT04460742/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/42/NCT04460742/ICF_001.pdf